CLINICAL TRIAL: NCT05242692
Title: The Effects of Subanesthetic S-ketamine on Postoperative Delirium and Cognitive Function in the Elderly Undergoing Non-cardiac Thoracic Surgery: a Protocol for Randomized, Double-blinded, placebo-and Positive-controlled, Non-inferiority Trial
Brief Title: The Effects of Subanesthetic S-ketamine on Postoperative Delirium and Cognitive Function in the Elderly Undergoing Non-cardiac Thoracic Surgery
Acronym: SKED
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ATHGuangzhou
Record Dates: First submitted 2021-12-23; First posted 2022-02-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Delirium; Elderly Patients
Keywords: Postoperative delirium; S-ketamine; Dexmedetomidine; elderly patients
MeSH Terms: conditions — Emergence Delirium | interventions — Esketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The labeled "Study medication" syringes (50ml) in identical appearance, and the infusion regimen formulated by the pharmacist based on the randomization, will be distributed to the attending anesthesiologists responsible for anesthetic management as soon as the research team informs the central pharmacy about the patient heading for surgery. To avoid anesthesiologists' speculation about the randomized assignment, the study drugs will be infused at a similar rate. The anesthesiologists, the patients, the investigators responsible for follow-up, and the statisticians are all masked to randomized allocations until the final statistical analyses are completed. The blindness will be unmasked by the primary investigator in a medical emergency including deterioration of patient's condition intraoperatively or adverse events postoperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-ketamine (Experimental): S-ketamine (50 mg, 2 ml) is diluted to 50 ml (1 mg/ml) with 48 ml normal saline;
  Interventions: Drug: S-ketamine
- Dexmedetomidine (Active Comparator): Dexmedetomidine (200 ug, 2 ml) is diluted to 100 ml (2 ug/ml) with 98 ml normal saline;
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: S-ketamine — Loading dose: 0.25mg/kg in 10 minutes Maintenance dose: 0.1mg/kg/h
  Arms: S-ketamine
Drug: Dexmedetomidine — Loading dose: 0.2 ug/kg in 10 minutes Maintenance dose: 0.2 ug/kg/h
  Arms: Dexmedetomidine

SUMMARY:
Postoperative delirium (POD) is a common and distressing complication after thoracic surgery. S-ketamine has neuroprotective properties as a dissociative anesthetic. Emerging literature has indicated that S-ketamine can reduce cognitive impairment in depressed patients. However, the role of S-ketamine in preventing postoperative delirium is still unknown. Therefore, this study aims to evaluate the effect of intraoperatively prophylactic S-ketamine compared to dexmedetomidine on the incidence of postoperative delirium in elderly patients undergoing non-cardiac thoracic surgery.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is a common and distressing complication after thoracic surgery. S-ketamine has neuroprotective properties as a dissociative anesthetic. Emerging literature has indicated that S-ketamine can reduce cognitive impairment in depressed patients. However, the role of S-ketamine in preventing postoperative delirium is still unknown. Therefore, this study aims to evaluate the effect of intraoperatively prophylactic S-ketamine compared to dexmedetomidine on the incidence of postoperative delirium in elderly patients undergoing non-cardiac thoracic surgery. This will be a randomized, double-blinded, placebo-and positive-controlled, non-inferiority trial that enrolls patients aged 60 or over undergoing thoracic surgery. The primary outcome will be the incidence of postoperative delirium within 4 days after surgery and assessed using a 3-minute Diagnostic Confusion Assessment Method (3D-CAM) twice a day. The main secondary outcomes will be the severity and duration of postoperative delirium. Other prespecified secondary outcomes will be the incidence of emergency delirium, postoperative pain, quality of sleep, cognitive function, and the plasm concentration of acetylcholine, brain-derived neurotrophic factor, and tumor necrosis factor.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or over
* Both genders
* American anesthesiologist association (ASA) physical status classificationⅠ-Ⅲ
* Diagnosed with lung, esophagus, or mediastinum disorders
* Undergoing open or video-assisted thoracic surgery including lobectomy, segmentectomy, pneumonectomy, esophagectomy, or resection of mediastinal tumor
* General anesthesia with one-lung ventilation (OLV) or bronchial blocker.
* An expected operation duration of 2 hours or more.
* Voluntarily participate in the trial and sign informed consent.

Exclusion Criteria:

* History of psychiatric disease or severe depression
* History of glaucoma or hyperthyroidism
* History of severe hepatic (Child-Pugh grade C) or renal (requirement for renal replacement therapy) disorder.
* Body mass index (BMI) greater 35 kg/m2
* Dementia history or baseline Mini-Mental State Examination (MMSE) score less than 23
* Severe audio-visual impairments, or inability to speak Mandarin or Cantonese precluding communication
* Sinus bradycardia (heart rate < 50 beats per minutes, bpm), sick sinus or Wolff- Parkinson-White syndromes, or Ⅱ degree atrioventricular block and over
* Poorly controlled hypertension (resting systolic blood pressure over 180 mm Hg, or resting diastolic blood pressure over 100 mm Hg)
* Allergic to dexmedetomidine, S-ketamine or any of their formulation ingredients;
* Taking sedatives, antidepressants or glucocorticoids
* Alcohol or drug abuser
* Life expectancy of less than 2 months due to extensive tumor metastasis.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Post-operative Delirium in 4 Days After Surgery | Within 4 days after surgery
  3-minute Diagnostic Confusion Assessment Method (3D-CAM)

SECONDARY OUTCOMES:
Severity of Delirium | Within 4 days after surgery
  Confusion Assessment Method- Severity (CAM-S, Mild-to-moderate delirium will be defined as a CAM-S score of 3 to 5, while severe delirium will be defined as a CAM-S score of 6 to 7)
Duration of postoperative delirium | Within 4 days after surgery
  Positive days of postoperative delirium

OTHER OUTCOMES:
Emergency delirium | From 30 minutes after the arrival in the post anesthesia care unit (PACU) until the time-point of PACU discharge, assessed up to 2 hours
  Richard Agitation-Sedation Scale (RASS) (RASS score ≥ 1 indicates emergency delirium, the higher scores mean a worse outcome.)
Pain severity | Within 2 days after surgery
  Numeric rating scale (NRS)0 = [no pain], 0 < NRS < 4 [mild pain], 4 ≤ NRS < 7 [moderate pain], 7 ≤ NRS <10 [severe pain], NRS = 10 [worst pain imaginable]
Quality of sleep | Within 4 days after surgery
  Numeric rating scale(0 = best-quality sleep, 10 = worst-quality sleep)
Cognitive function | On postoperative day 30
  Telephone interview for cognitive status-40 (TICS-40); A score below 21 will be defined as mild cognitive impairment, the higher scores mean a worse outcome.
Cognitive function | On postoperative day 90
  Telephone interview for cognitive status-40 (TICS-40); A score below 21 will be defined as mild cognitive impairment, the higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yihua Li, PhD, Study Chair — Cancer hospital and institute of Guangzhou medical university
Locations (1):
- Cancer hospital and institute of Guangzhou medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei W, Zhang A, Liu L, Zheng X, Tang C, Zhou M, Gu Y, Yao Y. Effects of subanaesthetic S-ketamine on postoperative delirium and cognitive function in elderly patients undergoing non-cardiac thoracic surgery: a protocol for a randomised, double-blinded, placebo-controlled and positive-controlled, non-inferiority trial (SKED trial). BMJ Open. 2022 Aug 1;12(8):e061535. doi: 10.1136/bmjopen-2022-061535. PMID 35914911

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT05242692/Prot_SAP_001.pdf